CLINICAL TRIAL: NCT00002260
Title: An Open-Label, Crossover Study to Assess the Effect of Food on the Oral Bioavailability and Pharmacokinetic Profile of 3'-Deoxy-3'-Fluorothymidine (FLT) in Asymptomatic Human Immunodeficiency Virus (HIV)-Infected Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lederle Laboratories (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 054C; 81-3
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-03

CONDITIONS: HIV Infections
Keywords: Biological Availability; alovudine; Food
MeSH Terms: conditions — HIV Infections | interventions — alovudine

INTERVENTIONS:
Drug: Alovudine

SUMMARY:
To characterize the pharmacokinetics of orally administered FLT (in a liquid formulation) after single doses in both the fed and fasting states; to assess the effect of food on the oral bioavailability of FLT

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Positive ELISA test confirmed by Western blot analysis.
* Asymptomatic.
* Willing to sign an informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Oral candida infection documented by morphology or by a response to antifungal therapy within two months prior to study entry.
* Oral hairy leukoplakia at any time prior to entry.
* Temperature > 37.8 C.
* Any malignancy other than cutaneous basal cell carcinoma or cervical carcinoma in situ.
* Significant chronic underlying medical illness which would prevent continuous participation in this clinical trial.
* Unwilling to sign an informed consent.
* Zidovudine induced hematological toxicity.

Prior Medication:

Excluded:

* Therapy with antiretroviral drugs or immunomodulators within seven days before entry.
* Therapy with any investigational drug during the preceding 30 days.

Patients may not have:

* Oral candida infection documented by morphology or by a response to antifungal therapy within two months prior to study entry.
* Oral hairy leukoplakia at any time prior to entry.
* Temperature > 37.8 C.
* Any malignancy other than cutaneous basal cell carcinoma or cervical carcinoma in situ.
* Significant chronic underlying medical illness which would prevent continuous participation in this clinical trial.
* Unwilling to sign an informed consent.
* Zidovudine induced hematological toxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Hosp, Baltimore, Maryland, United States